CLINICAL TRIAL: NCT00714545
Title: Intracoronary Brachytherapy for Recurrent Restenosis After Multiple Drug-Eluting Stents. Short Title: Scripps V
Brief Title: SCRIPPS V: Intracoronary Brachytherapy for Recurrent Restenosis After Multiple Drug-Eluting Stents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, Paul S Teirstein, MD, Director, Scripps Cardiovascular Institute, Scripps Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 004408
Record Dates: First submitted 2008-07-09; First posted 2008-07-14 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Coronary Artery Disease; Coronary Restenosis
Keywords: Coronary Artery Disease; Coronary Restenosis; Brachytherapy
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- prospective study (No Intervention): This study is a prospective study of patients treated at Scripps Clinic with intracoronary brachytherapy for recurrent restenosis within drug-eluting stents. Beta irradiation with a 40-mm strontium/yttrium-90 source. No placebo will be used in this trial.
  Interventions: Radiation: Intracoronary brachytherapy

INTERVENTIONS:
Radiation: Intracoronary brachytherapy — Beta irradiation with a 40-mm strontium/lytrium-90 source

SUMMARY:
This study is a prospective study of patients treated at Scripps Clinic with intracoronary brachytherapy for recurrent restenosis within drug eluting stents.

DETAILED DESCRIPTION:
This is an investigator-initiated protocol examining the effectiveness of intracoronary brachytherapy using the Novoste beta-emitting catheter for recurrent stenosis after treatment with multiple drug-eluting stents. While intracoronary brachytherapy has been used for this purpose by clinicians for some time, data supporting this clinical decision-making is lacking.

Currently, when cardiologists find restenosis after implanting a drug-eluting stent, they often place a stent that elutes a different drug within that stent. If a patient presents with restenosis in the segment that has already been treated with both sirolimus and paclitaxel-eluting stents, further options are limited. Intracoronary brachytherapy is often used in this scenario, but the efficacy of this approach has not been well studied. The investigators recently reviewed the clinical outcomes of five patients who underwent intracoronary radiation after drug-eluting stents. They discovered only one episode of target vessel revascularization and no episodes of stent thrombosis. While this sample is small, investigators believe that a prospective study will provide important information regarding this approach.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Eligible for percutaneous coronary intervention.
3. Target lesion with recurrent restenosis (>50% by visual estimate) previously treated with any 2 or more combination of DES stents.
4. Signs or symptoms of ischemia attributable to the target lesion, or stenosis > 50% by visual estimation of the lesion during angiography.
5. Target lesion is located within a native coronary artery or bypass graft.
6. Be reliable, cooperative and willing to comply with all protocol-specified procedures and follow-up.
7. Able to understand and sign informed consent.

Exclusion Criteria:

1. Confirmed pregnancy at the time of index PCI.
2. Has known allergies to aspirin, and to both clopidogrel (Plavix ®) and ticlopidine (Ticlid ®).
3. Has known allergies or contraindication to heparin and Bivalirudin (Angiomax ®).
4. Has a significant medical condition which in the investigator's opinion may interfere with the patient's optimal participation in the study.
5. Any serious disease condition with life expectancy of less than 1 year.
6. Unsuccessful coronary revascularization procedure (residual stenosis > 30%).
7. Angiographic evidence of thrombus.
8. No Previous intracoronary radiation to the target artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To determine the safety and efficacy of intracoronary brachytherapy for the treatment of recurrent restenosis within drug-eluting stents. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Paul S. Teirstein, MD, Principal Investigator — Scripps Clinic
Locations (1):
- Scripps Green Hospital/Scripps Clinic, La Jolla, California, United States